CLINICAL TRIAL: NCT00628485
Title: BION Stimulation to Improve Swallowing Function After Radical Head-neck Surgery and Follow-up Chemoradiation Therapy
Brief Title: BION Treatment of Dysphagia After Radical Head-Neck Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Gerald E. Loeb, M.D., Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BT9
Record Dates: First submitted 2008-02-25; First posted 2008-03-05 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Dysphagia
Keywords: swallowing function; neuromuscular stimulator
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low Stimulation (Experimental): The first group will have a stimulation paradigm employing low-frequency (1-5 pps), supramaximal "twitch" stimulation.
  Interventions: Device: BION
- High Stimulation (Experimental): The second group will have a "High Stimulation" paradigm at a frequency that produces strong, fused contractions (20-30pps) for a total of 1h/d, also in two spaced sessions.
  Interventions: Device: BION
- Control Group (Placebo Comparator): A third group of experimental subjects will have a standardized program of voluntary swallowing exercises.
  Interventions: Device: BION

INTERVENTIONS:
Device: BION — The second group will have a "High Stimulation" paradigm at a frequency that produces strong, fused contractions (20-30pps) for a total of 1h/d, also in two spaced sessions. Stimulation intensity will be adjusted to produce the strongest contractions that are tolerated.
  Arms: High Stimulation
Device: BION — The first group will have a stimulation paradigm employing low-frequency (1-5 pps), supramaximal "twitch" stimulation. The period of the stimulation will probably be short for the first sessions as the muscles gain strength and fatigue resistance, but will eventually be 60 minutes per day in two spaced sessions of about 30 minutes each.
  Arms: Low Stimulation
Device: BION — A third group of experimental subjects will have a standardized program of voluntary swallowing exercises. Their BIONs will not be activated until they have worsening of dysphagia, and thus are considered to have failed conventional therapy.
  Arms: Control Group

SUMMARY:
The primary goal of the proposed study is to improve the long-term swallowing capabilities of subjects undergoing radical or modified radical neck surgeries followed by chemoradiation therapy (CRT), by more selective stimulation of the swallowing muscles using implanted microstimulators called BIONs.

DETAILED DESCRIPTION:
Disseminated head and neck cancer is a serious, often life-threatening medical problem that requires immediate and heroic therapeutic intervention. Treatment typically begins with extensive surgery followed as soon as possible by an intense series of radiation and chemotherapy treatments. Typically the patient has recovered sufficiently from the surgery by 2-4 weeks to withstand the new assaults that will result from chemoradiation therapy (CRT), which kills cancer cells, but also causes muscle atrophy and scarring that can permanently ruin the swallowing apparatus. Thus, the majority of patients who undergo CRT develop severe swallowing problems, called dysphagia, that typically becomes worse by about 3-4 weeks following the beginning of CRT. In anticipation of all of these problems, subjects have a tube placed in the stomach (gastrostomy tube) so that they can be fed through the tube in the immediate postoperative period when the incision is fragile and when dysphagia develops during CRT. Clearly the management of dysphagia during CRT is of primary importance to the prognosis of the patient. Recent studies have shown that electrical activation of swallowing muscles during and after CRT can improve the prognosis by reducing dysphagia, but currently available technology requires the current to be applied transcutaneously. Thus, large electrical currents must be applied to the damaged skin, and the electrical stimulation that results is uncomfortable, diffuse and uncontrolled. It is difficult with this approach to stimulate the deepest muscles that are the preferred targets for the stimulation. The primary goal of the proposed study is to improve the long-term swallowing capabilities of subjects undergoing radical or modified radical neck surgeries followed by CRT, by more selective stimulation of the swallowing muscles using implanted microstimulators called BIONs. The mechanism of the electrical stimulation is thought to be the same as that for other rehabilitative approaches to muscle, i.e.,to help maintain strength and mobility of these muscles during the post-operative treatment period when the muscles are not being used and are particularly vulnerable to scarring and atrophy.

Two different paradigms of stimulation will be employed in order to compare and gain insight into the mechanisms involved in the remediation. This study also presents the opportunity to examine directly the changes in muscle produced by stimulation. Thus, a secondary research goal of the study that takes advantage of the opportunity presented by this intervention is to gain insight into the cellular changes that are thought to underlie the effects of radiation and subsequent electrical stimulation. By implanting these devices at the time of the neck surgeries, it is possible to target the nerves that supply specific muscles and thus ensure the excitation of specific muscles using current strengths much lower than those required with transcutaneous stimulation.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has Stage 3-4 cancer of the oral cavity or oropharynx with a primary tumor size of 1-6 cm (T1-T3) and neck lymph node metastases.
2. Subject is above 18 years old.
3. Attending physician considers the subject to be an appropriate candidate for surgery and chemoradiation therapy.
4. Subject is mentally capable of understanding the goals and the application of therapy or whenever in doubt, is able to pass the Minimental State (MMSE) test.
5. Subject is able to apply the therapy without help or with the help of a caregiver.
6. Subject is willing and capable of giving informed consent.
7. Subject is willing and capable of traveling to testing center at the necessary points in the schedule of testing.

Exclusion Criteria:

1. Subject is pregnant, nursing, or planning to become pregnant in the next 12 months.
2. Subject has an electronic implant (e.g. cardiac pacemaker, etc.).
3. Subject has large metallic implant (e.g. skull plates) in the head or neck region (small metal implants, such as bone screws, metal sutures or dental parts are acceptable).
4. Subject has had previous surgery or disease of the upper esophageal tract or vocal structures that have changed the normal anatomical relationships of the epiglottal region, making swallowing abnormal, or have damaged the nerves of the target muscles that control swallowing, making it difficult to stimulate the swallowing muscles effectively.
5. Subject has an active immunosuppressive disorder such as AIDS that may result in muscle wasting, or has a neurological injury or disease that affects the function of the nerves or neuromuscular endplates in the throat, such as myasthenia gravis or multiple sclerosis. The subject has a significant concurrent or recently diagnosed (less than 3 months) medical condition that, in the opinion of the medical investigator, could affect the ability of the patient to tolerate or complete the study. Such conditions might include a second malignancy, heart disease or stroke.
6. Subject has a major psychological disorder, such as poorly controlled schizophrenia or paranoia, that may affect the clinical interactions with the subject or result in poor compliance with the therapy.
7. Subject has a significant respiratory problem such as asthma or chronic obstructive lung disease requiring regular use of inhaled or systemic corticosteroids. Subject has a tracheostomy or has had previous surgery on the trachea that has damaged the swallowing muscles or made inhalation of swallowed food more likely.
8. Subject is currently enrolled in another investigational study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2007-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
swallowing function | prior surgery, 2w post surgery, end of radiation recovery, end of rehab

SECONDARY OUTCOMES:
blood test, ease of swallowing questionnaire | prior surgery, 2w post surgery, end of radiation recovery, end of rahab

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Loeb, MD, Principal Investigator — University of Southern California
Locations (1):
- USC University Hospitals, Los Angeles, California, United States